CLINICAL TRIAL: NCT02023905
Title: PI3K/mTOR Pathway Activation Selected Phase II Study of Everolimus (RAD001) With and Without Temozolomide in the Treatment of Adult Patients With Supratentorial Low-Grade Glioma
Brief Title: Everolimus With and Without Temozolomide in Adult Low Grade Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Novartis-CRAD001CUS225T; 131012 (Other: University of California, San Francisco); NCI-2014-00749 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: Low Grade Glioma; World Health Organization (WHO) Grade II Astrocytomas; Oligodendrogliomas; Mixed Oligoastrocytomas
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Everolimus; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Everolimus (Experimental): If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If activation is present, patients will be treated with single-agent everolimus at 10 mg daily continuously for up to 24 cycles, after which patients will be followed with interval MRIs until progression.
  Interventions: Drug: Everolimus
- Arm 2: Everolimus and Temozolomide (Experimental): If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If activation is not present, patients will be treated with combined everolimus and Temozolomide (TMZ). Everolimus will be given at 10 mg daily continuously for up to 24 cycles, and Temozolomide will be dosed initially at 150 mg/m^2 per day for 5 days out of a 28-day cycle for up to 12 cycles, after which patients will be followed with interval MRIs until progression.
  Interventions: Drug: Everolimus; Drug: Temozolomide
- Arm 3: Everolimus (1p/19q co-deletion present) (Experimental): If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If 1p/19q co-deletion is present, patients will be treated with single-agent everolimus at 10 mg daily continuously for up to 24 cycles, after which patients will be followed with interval MRIs until progression.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — everolimus at 10 mg daily continuously
  Other Names: RAD001, Afinitor
Drug: Temozolomide — Temozolomide will be dosed initially at 150 mg/m2/day for 5 days out of a 28-day cycle. TMZ will be stopped after 12 cycles
  Other Names: Temodar, TMZ
  Arms: Arm 2: Everolimus and Temozolomide

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, everolimus (RAD001, also known as Afinitor®) alone or with temozolomide has on the patient and the patient's low-grade glioma. Everolimus is being investigated as an anticancer agent based on its potential to prevent tumor cells from growing and multiplying. Specifically, there is a protein called mTOR that we think helps many tumors to grow, and everolimus blocks the effect of mTOR. Temozolomide is also an anticancer agent that prevents tumor cells from growing and multiplying.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Arm 1: To assess progression-free survival in patients with previously untreated alpha-thalassemia/mental retardation, X-linked (ATRX) lost and/or 1p/19q intact, phosphatidylinositol 3-kinase (PI3K)/Mechanistic target of rapamycin (mTOR) pathway-activated low grade-glioma (LGG) treated with everolimus.

Arm 2: To assess progression-free survival in patients with previously untreated ATRX lost and/or 1p/19q intact, PI3K/mTOR pathway-non-activated LGG treated with everolimus and TMZ.

Arm 3: To assess progression-free survival in patients with previously untreated ATRX intact and/or 1p/19q co-deleted LGG treated with everolimus.

SECONDARY OBJECTIVES:

1. To assess overall and progression-free survival distributions (Arms 1, 2 & 3).
2. To assess the objective response rate to treatment (Arms 1, 2 & 3).
3. To further delineate the safety profile of the combination of everolimus and TMZ (Arm 2)
4. To assess whether treatment (Arms 1, 2 & 3) provides clinical benefit by reducing seizure frequency

EXPLORATORY OBJECTIVES

1. Pending adequate funding, to assess the ability of metabolic and physiologic imaging parameters such as magnetic resonance (MR) spectroscopy, perfusion-weighted imaging, and diffusion-weighted imaging to predict clinically relevant endpoints such as time to progression and survival.
2. To assess for an association between the presence/absence of clonal or subclonal genetic mutations in the PI3K pathway and Median progression-free survival (PFS), Objective Response Rate (ORR), phosphatase and tensin homolog (PTEN) gene methylation, and the immunohistochemical measurements of the PI3K pathway activation in patients treated with everolimus or TMZ and everolimus.
3. To longitudinally assess quality of life (QoL) in low-grade glioma patients over the course of treatment with everolimus (Arms 1 & 3).

OUTLINE:

Patients will be assigned to one of 3 treatment arms based on two characteristics of their tumor, called "1p/19q" (this is a test of the tumor chromosomes) and "p-PRAS40" (this is a test of a pathway in the tumor called mTOR). If the patient's tumor is 1p/19q intact and the phosphorylation of proline-rich Ak strain transforming (AKT) substrate of 40 kDa, encoded by the gene AKT1S1 (p-PRAS40) positive, the patient will be assigned to Treatment Arm 1. If the patient's tumor is 1p/19q intact and p-PRAS40 negative, the patient will be assigned to Treatment Arm 2. If the patient's tumor is 1p/19q co-deleted, regardless of the p-PRAS40 result, the patient will be assigned to Treatment Arm 3.

All patients will be observed for safety for 30 days following the last dose of everolimus. After completion of study treatment, patients whose tumors have not progressed will be followed with interval MRIs for an additional 2 years, and thereafter as per the discretion of the managing physician. Patients off protocol therapy will continue to be followed for survival only.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Karnofsky performance scale score (KPS) >= 60
* Adequate bone marrow function as shown by: Absolute Neutrophil Count (ANC) >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, hemoglobin >= 9.0 g/dL;
* Adequate liver function as shown by: Total serum bilirubin ≤ 2.0 mg/dL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5x upper limit of normal (ULN), International Normalized Ratio (INR) <= 2;
* Adequate renal function: serum creatinine <=1.5 x ULN;
* Fasting serum cholesterol <= 300 mg/dL OR <= 7.75 mmol/L AND fasting triglycerides <= 2.5x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication with confirmed reduction of lab values to within eligibility parameters;
* Signed informed consent prior to any screening procedures
* Histologically proven supratentorial low-grade glioma at initial diagnosis; pathology must have been reviewed by University of California, San Francisco (UCSF) neuropathology. Eligible low-grade gliomas include: astrocytoma, oligodendroglioma and mixed oligoastrocytoma. Pilocytic astrocytomas are excluded.
* Patient's tumor must have documentation of the presence of an Isocitrate dehydrogenase 1 (IDH1) and/or Isocitrate dehydrogenase 2 (IDH2) mutation of any type.
* Results of 1p/19q chromosomal status and p-PRAS40 testing must be available to permit treatment selection.
* Evaluable disease
* Must begin treatment within 120 days of surgical procedure

Exclusion Criteria:

* No prior tumor treatment except for surgery at diagnosis, and must have adequately recovered from surgery
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus) or to temozolomide
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus or temozolomide
* Uncontrolled diabetes mellitus as defined by HbA1c > 8.0% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary;
* Any severe and/or uncontrolled medical conditions such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease; symptomatic congestive heart failure of New York heart Association Class III or IV; active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus(HBV-DNA and/or positive Hepatitis B Surface Antigen (HbsAg), quantifiable hepatitis C virus (HCV-RNA); known severely impaired lung function (spirometry and Diffusing capacity of the lungs for carbon monoxide (DLCO) 50% or less of normal and O2 saturation 88% or less at rest on room air); active, bleeding diathesis;
* Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed, and treatment with low dose Decadron (<= 3mg daily) is allowed;
* Known history of HIV seropositivity;
* Positive serological test results for hepatitis B
* Positive serological test result for hepatitis C
* Recipients of live attenuated vaccines within 1 week of start of treatment and during the study. Avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines;
* History of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uterus, or breast, unless the patient has been disease free for >= 3 years;
* History of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study;
* Currently part of or have participated in any clinical investigation with an investigational therapeutic drug within 1 month prior to dosing;
* Pregnant or nursing (lactating) women;
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, who are not willing to use adequate methods of contraception during the study and for 8 weeks after the end of treatment.
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Abstract: Neuro Oncol. 2019 Nov; 21(Suppl 6): vi22-vi23 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6846978/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Everolimus: If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the phosphatidylinositol 3-kinase (PI3K)
  /Mechanistic target of rapamycin (mTOR) pathway. If activation is present, patients will be treated with single-agent everolimus at 10 mg daily continuously for up to 24 cycles.
- Arm 2: Everolimus and Temozolomide: If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If activation is not present, patients will be treated with combined everolimus and temozolomide (TMZ). Everolimus will be given at 10 mg daily continuously for up to 24 cycles, and Temozolomide will be dosed initially at 150 mg/m^2 per day for 5 days out of a 28-day cycle for up to 12 cycles.
- Arm 3: Everolimus (1p/19q Co-deletion Present): If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If 1p/19q co-deletion is present, patients will be treated with single-agent everolimus at 10 mg daily continuously for up to 24 cycles.
Period: Overall Study
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
Started | 16 | 2 | 9
Completed | 16 | 2 (One participant went off treatment after a few days of beginning therapy due to adverse events, but is included in the efficacy analysis as completed under the intent-to-treat (ITT) model.) | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Everolimus: If the tumor is 1p/19q intact, then patients will be further selected by whether or not their tumor demonstrates activation of the PI3K/mTOR pathway. If activation is present, patients will be treated with single-agent everolimus at 10 mg daily continuously for up to 24 cycles.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present) | Total
Number analyzed (Participants) | 16 | 2 | 9 | 27
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 6 | 1 | 3 | 10
  30-39 years old | 4 | 1 | 1 | 6
  40-49 years old | 2 | 0 | 1 | 3
  50-59 years old | 2 | 0 | 4 | 6
  60-69 years old | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 12 | 0 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 15 | 1 | 8 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 13 | 0 | 8 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 2 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Rate (PFS) (Arms 1 and 2)
Description: Participants will be analyzed based on intention to treat using the Response Assessment in Neuro-Oncology (RANO) criteria for progression. Based on RANO criteria, a responder is defined using both radiographic and clinical criteria. Complete response (CR) or Partial Response (PR) will be first assessed by radiographic changes as determined by an improvement of the bi-dimensional evaluation of the tumor size. In addition, changes in neurologic function and steroid use will be considered. Analyses will be performed after all enrolled participants in arm 1 or arm 2 have completed 33 months on study, or whenever the progression status of all participants has been established, whichever comes first. Kaplan-Meier estimates and the associated 95% confidence intervals (CI) will be calculated for the 33-month PFS separately for the two arms.
Time Frame: Up to 33 Months
Population: One participant in Arm 2 went off treatment after only a few days of beginning therapy but was included in the analysis as part of the ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide
Number analyzed (Participants) | 16 | 2
percentage of participants | 31 [15.1 to 64.6] | NA [NA to NA] — There were insufficient number of events so an estimate and confidence interval could not be calculated.

2. Primary Outcome: Progression-Free Survival Rate (PFS) (Arm 3)
Description: Participants will be analyzed based on intention to treat using the Response Assessment in Neuro-Oncology (RANO) criteria for progression. Based on RANO criteria, a responder is defined using both radiographic and clinical criteria. Complete response (CR) or Partial Response (PR) will be first assessed by radiographic changes as determined by an improvement of the bi-dimensional evaluation of the tumor size. In addition, changes in neurologic function and steroid use will be considered. Analyses will be performed after all participants enrolled in arm 3 have completed 38 months on study, or whenever the progression status of all participants has been established, whichever comes first. Kaplan-Meier estimates and the associated 95% CIs will be calculated for the 38-month PFS.
Time Frame: Up to 38 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 3: Everolimus (1p/19q Co-deletion Present)
Number analyzed (Participants) | 9
percentage of participants | 55.5 [31 to 99.7]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Participants will be analyzed based on an intention to treat model. PFS is defined as the time from first objective response to the time of disease progression or death using the Response Assessment in Neuro-Oncology (RANO) criteria to determine progression. If the participant does not have an event of disease progression or recurrence nor has the patient died, the participant's data will be censored at the date of last contact with the patient. Kaplan-Meier estimates and the associated 95% CIs will be calculated.
Time Frame: Up to 84 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
Number analyzed (Participants) | 16 | 2 | 9
months | 25.8 [19.2 to NA] — The upper range of the confidence interval was calculated to be infinity. | NA [NA to NA] — There were insufficient number of events so an estimate and confidence interval could not be calculated. | 43.6 [19.4 to NA] — The upper range of the confidence interval was calculated to be infinity.

4. Secondary Outcome: Overall Survival Rate (OS)
Description: Participants will be analyzed based on an intention to treat model. Overall survival is defined as the first day of treatment until death or study completion, whichever comes first. Kaplan-Meier estimates and the associated 95% CIs will be calculated by treatment arm.
Time Frame: Up to 84 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
Number analyzed (Participants) | 16 | 2 | 9
percentage of participants | NA [86.8 to NA] — There were insufficient number of events (2) so an estimate could not be calculated and the upper range of the confidence interval was calculated to be infinity. | NA [NA to NA] — There were insufficient number of events so an estimate and confidence interval could not be calculated. | NA [NA to NA] — There were insufficient number of events (0) so an estimate and confidence interval could not be calculated.

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Overall response rate (ORR) is the percentage of patients who achieved a best response of complete response (CR) or partial response (PR) out of all assigned patients. Based on the best objective status as assessed by the Response Assessment in Neuro-Oncology (RANO) criteria. Using RANO criteria, a responder is defined by radiographic and clinical criteria. Complete response or PR will be first assessed by radiographic changes as determined by an improvement of the bi-dimensional evaluation of the tumor size. In addition, changes in neurologic function and steroid use will be considered. The point estimate and the associated 2-sided 95% CI for the response rate separately for the three arms.
Time Frame: Up to 36 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
Number analyzed (Participants) | 16 | 2 | 9
percentage of participants | 0 [0 to 19.4] | NA [NA to NA] — There were insufficient numbers of participants with events so the ORR and confidence interval could not be calculated | 11 [5.7 to 43.5]

6. Secondary Outcome: Rate of Reduction in Seizures
Description: To assess the reduction in seizure rate the investigator will compare the seizure rate on study to that experienced one month prior to enrolling in the study. The RANO low grade gliomas (LGG) guideline will be used to assess reduction of seizures, which calls a 50% or more reduction number of monthly seizures an 'improvement'; a 50% or more increase a worsening'; and anything less than 50% in either direction a 'stable seizure rate'.
Time Frame: Up to 36 Months
Population: One participant in Arm 2 went off treatment after only a few days of beginning therapy, so monthly seizure data could not be collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
Number analyzed (Participants) | 16 | 1 | 9
percentage of participants | 25 [8.9 to 53.2] | NA [NA to NA] — Rate and confidence interval could not be calculated for single participant | 50 [21.5 to 78.5]

ADVERSE EVENTS:
Time Frame: Up to 84 months
Arm/Group | Arm 1: Everolimus | Arm 2: Everolimus and Temozolomide | Arm 3: Everolimus (1p/19q Co-deletion Present)
All-Cause Mortality (participants affected / at risk) | 2/16 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/2 | 3/9
Other Adverse Events (participants affected / at risk) | 12/16 | 1/2 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Everolimus (N=16) | Arm 2: Everolimus and Temozolomide (N=2) | Arm 3: Everolimus (1p/19q Co-deletion Present) (N=9)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Uterine Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Everolimus (N=16) | Arm 2: Everolimus and Temozolomide (N=2) | Arm 3: Everolimus (1p/19q Co-deletion Present) (N=9)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 6 (19) | 1 (5) | 6 (24)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 1 (1) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (8) | 0 (0) | 5 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (7) | 1 (1) | 3 (3)
General disorders and administration site conditions - Other (General disorders) | 2 (2) | 1 (1) | 2 (3)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 3 (4) | 0 (0) | 2 (8)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 2 (8)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Memory Impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 1 (5) | 4 (17)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0) | 5 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (4) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Neck pain (Investigations) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was closed prematurely due to slow accrual and loss of drug support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02023905/Prot_SAP_000.pdf